CLINICAL TRIAL: NCT05573802
Title: A Phase 1/2, Dose and Schedule Evaluation Study to Investigate the Safety and Clinical Activity of Belantamab Mafodotin Administrated in Combination With Lenalidomide, Dexamethasone and Nirogacestat in Patients With Transplant Ineligible Newly Diagnosed Multiple Myeloma
Brief Title: A Study to Investigate Safety and Clinical Activity of Belantamab Mafodotin in Combination With Lenalidomide, Dexamethasone and Nirogacestat in Patients With Transplant Ineligible Newly Diagnosed Multiple Myeloma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hellenic Society of Hematology (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: EAE128
Record Dates: First submitted 2022-10-06; First posted 2022-10-10 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Multiple Myeloma; Neoplasms; Neoplasm, Plasma Cell; Gammopathy, Monoclonal; Paraproteinemias; Blood Protein Disorders; Haematologic Disease; Corneal Disease
MeSH Terms: conditions — Multiple Myeloma; Neoplasms; Neoplasms, Plasma Cell; Paraproteinemias; Blood Protein Disorders; Hematologic Diseases; Corneal Diseases | interventions — Lenalidomide; Dexamethasone; nirogacestat

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Part 1 : Dose finding (Experimental): Belantamab mafodotin will be administered as a combination therapy as a calculated dose on Day 1 of every other 28-day cycle.
  Belantamab mafodotin starting dose:
  • 1.4 mg/kg Q8W (i.e., on Day 1 of every other 28-day cycle)
  * Dose Level +1: 1.9 mg/kg Q8W
  * Dose Level -1: 1.0 mg/kg Q8W
  * Dose Level -2: 1.0 mg/kg Q12W
  Lenalidomide: 25 mg/d on day 1-21 of every 28-day cycle.
  Dexamethasone: 40 mg/d on days 1, 8, 15, 22 of every 28-day cycle in participants < 75 years; 20 mg/d on days 1, 8, 15, 22 of every 28-day cycle in participants ≥ 75 years
  Nirogacestat: 100 mg twice a day (BID) starting on day -3 and then each day of every other 28-day cycle (i.e., to be given only on cycles where belantamab mafodotin is administered).
  Interventions: Drug: Belantamab Mafodotin-Blmf; Drug: Lenalidomide; Drug: Dexamethasone; Drug: Nirogacestat

INTERVENTIONS:
Drug: Belantamab Mafodotin-Blmf — Blmf will be available as 100 mg/vial in single-use vial for reconstitution, supplied as lyophilized powder. Blmf will be delivered as IV solution over at least 30 minutes.
Drug: Lenalidomide — Lenalidomide will be administered per os.
Drug: Dexamethasone — Dexamethasone will be administered intravenously or per os.
Drug: Nirogacestat — Nirogacestat will be administrated each day for all subsequent cycles were Blmf is also administrated.

SUMMARY:
This is a phase 1/2, open-label study designed to assess the safety and clinical activity of different belantamab mafodotin doses in combination with lenalidomide, dexamethasone and nirogacestat in patients with transplant ineligible newly diagnosed multiple myeloma.

This will be a 2-part study. In part 1 participants will be enrolled in one cohort to receive belantamab mafodotin in combination with lenalidomide, dexamethasone and nirogacestat and will determine the recommended phase 2 dose (RP2D) to be further evaluated for safety and clinical activity in the dose expansion cohort. The RP2D dose will be used in future studies in the transplant-ineligible newly diagnosed multiple myeloma (NDMM) setting. In the dose expansion phase (Part 2) an expansion cohort will be treated with the RP2D. The expansion cohort will randomize participants (1:1) in two groups to evaluate two alternate dose modification guidelines for corneal AEs. Part 2 of the study will also evaluate an alternative dose modification guideline for corneal adverse events (AEs).

Overall, approximately 36 participants will be enrolled in the study. Participant follow-up will continue up to 3 years after the last participant is enrolled (follow-up period range: 3-4 years). The estimated accrual period will be 12 months, corresponding to an approximate total study duration of 4 years.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be >18 years of age
2. Monoclonal plasma cells in the bone marrow (BM) ≥10% or presence of a biopsy proven plasmacytoma and documented Multiple Myeloma (MM) satisfying at least one of the calcium, renal, anemia, bone (CRAB) criteria or biomarkers of malignancy criteria:

   CRAB criteria:

   i. Hypercalcemia: serum calcium >0.25 mmol/L (>1 mg/dL) higher than upper limit of normal (ULN) or >2.75 mmol/L (>11 mg/dL).

   ii. Renal insufficiency: creatinine clearance (CrCI) <40mL/min or serum creatinine >177 μmol/L (>2 mg/dL).

   iii. Anemia: hemoglobin >2 g/dL below the lower limit of normal or hemoglobin <10 g/dL.

   iv. Bone lesions: one or more osteolytic lesions on skeletal radiography, Computed tomography (CT), or Positron emission tomography (PET-CT).

   Biomarkers of Malignancy:
   1. Clonal BM plasma cell percentage ≥60%.
   2. Involved: uninvolved serum free light chain (sFLC) ratio ≥100.
   3. More than 1 focal lesion on magnetic resonance imaging (MRI) studies.
3. Must have at least ONE aspect of measurable disease, defined as one of the following:

   * Urine M-protein excretion ≥200 mg/24 hrs (≥0.2 g/24 hrs), or
   * Serum M-protein concentration ≥0.5 g/dL (≥5.0 g/L), or
   * Serum FLC assay: involved FLC level ≥10 mg/dL (≥100 mg/L) and an abnormal serum FLC ratio (<0.26 or >1.65).
4. Not a candidate for high-dose chemotherapy with autologous stem cell transplantation due to presence of significant comorbid condition(s), such as cardiac, pulmonary or other major organ dysfunction that are likely to have a negative impact on tolerability of high dose chemotherapy with stem cell transplantation. The patients will be assessed with the IMWG frailty index, a scoring system based on age, comorbidities, and cognitive and physical conditions, which is recommended by the European Society for Medical Oncology (ESMO) guidelines. Patients with International Myeloma Working Group (IMWG) frailty index score 1 or 2 will be considered transplant ineligible. The reason(s) for transplant ineligibility will be collected in the case report forms (CRFs).
5. Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0-2.
6. Adequate organ system function as defined by the below laboratory assessments. Hematologic

   * Absolute neutrophil count (ANC) ≥1.25 X 10^9/L; granulocyte colony-stimulating factor (G-CSF) use for the past 14 days is NOT allowed.
   * Hemoglobin ≥8.0 g/dL; transfusions are not permitted in the past 14 days prior to the assessment. Erythropoietin use is allowed.
   * Platelet count ≥50 x 10^9/L if the BM is >50% involved in myeloma. Otherwise, ≥75 x 10^9/L; transfusions or platelet stimulating agents are NOT allowed in the past 14 days prior to the assessment.

   Hepatic
   * Total bilirubin ≤1.5xULN (isolated bilirubin ≥1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
   * ALT ≤ 2.5xULN. Renal
   * Estimate glomerular filtration rate (eGFR) ≥30 mL/min/1.73 m2; calculated using the Modified Diet in Renal Disease (MDRD) formula.
   * Spot urine (albumin/creatinine ratio) <500 mg/g (56 mg/mmol) OR
   * Urine Dipstick: Negative trace; if ≥1+ only eligible if confirmed <500 mg/g [56 mg/mmol] by albumin/creatinine ratio (spot urine from first void).
7. Female participants: contraceptive use should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies:

   A female participant is eligible to participate if she is not pregnant or breastfeeding, and at least one of the following conditions applies:
   * Is not a woman of childbearing potential (WOCBP) defined as follows:
   * ≥ 45 years of age and has not had menses for > 1 year
   * Patients who have been amenorrhoeic for < 2 years without history of a hysterectomy and oophorectomy must have a follicle stimulating hormone value in the postmenopausal range upon screening evaluation
   * Post-hysterectomy, post-bilateral oophorectomy, or post-tubal ligation. Documented hysterectomy or oophorectomy must be confirmed with medical records of the actual procedure or confirmed by an ultrasound. Tubal ligation must be confirmed with medical records of the actual procedure.

   OR
   * Is a WOCBP and using two methods of reliable birth control (one method that is highly effective and one additional effective [barrier] method), beginning 4 weeks before initiating treatment with lenalidomide, during therapy, during dose interruptions and continuing for 4 weeks following discontinuation of lenalidomide treatment. WOCBP participants must use one method of reliable birth control that is highly effective for 4 months following discontinuation of belantamab mafodotin. WOCBP must also agree not to donate eggs (ova, oocytes) for the purpose of reproduction during treatment, during dose interruptions and for 28-days following the last dose of lenalidomide or 4 months following discontinuation of belantamab mafodotin treatment, whichever is longer.

   A WOCBP must have two negative pregnancy tests before therapy initiation. The first test should be performed within 10-14 days, and the second test within 24 hours before the start of lenalidomide therapy.

   The participant should not receive lenalidomide until the investigator has verified that the results of these pregnancy tests are negative. The investigator should evaluate the effectiveness of the contraceptive method in relation to the first dose of the study treatment. The investigator is responsible for a review of medical history, menstrual history, and recent sexual activity to decrease the risk for inclusion of a woman with a nearly undetected pregnancy.

   WOCBP is a female who:
   * has achieved menarche at some time point
   * has not undergone a hysterectomy or bilateral oophorectomy or
   * has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months).
8. Male participants: contraceptive use should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies:

   Male participants are eligible to participate if they agree to the following during the intervention period and until 28 days after the last dose of lenalidomide or 6 months after the last dose of belantamab mafodotin, whichever is longer, to allow for clearance of any altered sperm.
   * Refrain from donating sperm

   PLUS either:
   * Be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis) and agree to remain abstinent, OR
   * Must agree to use contraception/barrier as detailed below:

   Agree to use a male condom, even if they have undergone a successful vasectomy, and female partner to use an additional highly effective contraceptive method with a failure rate of <1% per year as when having sexual intercourse with a woman of childbearing potential (including pregnant females).
9. Participants must be able to understand the study procedures and agree to participate in the study by providing written informed consent.

Exclusion Criteria:

1. Prior systemic therapy for MM or Smoldering MM.

   * NOTE 1: An emergency course of steroids (defined as not greater than 40 mg of dexamethasone [or equivalent] per day for a maximum of 4 days [i.e., a total of 160 mg]) is permitted.
   * NOTE 2: Focal palliative radiation is permitted before enrollment, provided that: it occurred at least 2 weeks before the first dose of the study drug; the participant has recovered from radiation-related toxicities; and the participant did not require corticosteroid administration (for a longer period than that specified in NOTE 1 above) for radiation-induced AEs.
2. Peripheral neuropathy or neuropathic pain Grade 2 or higher, as defined by the National Cancer Institute Common Toxicity Criteria for AEs version 5.
3. Major surgery within 2 weeks before the first dose of the study drug.

   * NOTE 1: patients who underwent major surgery must be clinically stable to be enrolled in the study.
   * NOTE 2: major surgery shall be defined based on the Investigator's judgment according to the extent and complexity of the procedure, its pathophysiological consequences and consecutive clinical outcomes.
4. Presence of active renal condition (infection, requirement for dialysis or any other significant condition that could affect the participant's safety). Participants with isolated proteinuria resulting from MM are eligible, provided that they fulfil the other inclusion criteria.
5. Any serious and/or unstable pre-existing medical, psychiatric disorder, or other conditions (including laboratory abnormalities) that could interfere with the participant's safety, obtaining informed consent, or compliance with the study procedures.
6. Evidence of active mucosal or internal bleeding uncontrolled by local therapy and not explained by reversible coagulopathy.
7. Current active liver or biliary disease (except for Gilbert's syndrome or asymptomatic gallstones, or otherwise stable chronic liver disease as per the investigator's assessment).
8. Participants with previous or concurrent malignancies other than MM are excluded. Exceptions are surgically treated cervical carcinoma in situ or any other malignancy that has been considered medically stable for at least 2 years. The participant must not be receiving active therapy other than hormonal therapy for this disease.

   * NOTE: Participants with curatively treated non-melanoma skin cancer are allowed without a 2-year restriction.
9. Evidence of cardiovascular risk including any of the following:

   * Evidence of current clinically significant untreated arrhythmias, including clinically significant electrocardiogram (ECG) abnormalities, second degree (Mobitz Type II), or third degree atrioventricular (AV) block.
   * History of myocardial infarction, acute coronary syndromes (including unstable angina), coronary angioplasty, or stenting or bypass grafting within 3 months of screening.
10. Class III or IV heart failure as defined by the New York Heart Association functional classification system.
11. Uncontrolled hypertension.
12. Active infection requiring treatment.
13. Known HIV infection, unless the participant can meet all of the following criteria:

    * Established anti-retroviral therapy (ART) for at least 4 weeks and HIV viral load <400 copies/mL.
    * CD4+ T-cell (CD4+) count ≥350 cells/uL.
    * No history of AIDS-defining opportunistic infections within the last 12 months.

      * NOTE: consideration must be given to ART and prophylactic antimicrobials that may have a drug:drug interaction and/or overlapping toxicities with belantamab mafodotin or other combination products as relevant
14. Seropositivity for hepatitis B (defined by a positive test for hepatitis B surface antigen [HBsAg]).

    * NOTE 1: Participants with resolved infection (i.e., participants who are positive for antibodies to hepatitis B core antigen [antiHBc] or antibodies to hepatitis B surface antigen [antiHBs]) must be screened using real-time polymerase chain reaction (PCR). Those who are PCR positive will be excluded.
    * NOTE 2: presence of antiHBs indicating previous vaccination will not constitute an exclusion criterion.
15. Positive hepatitis C antibody test result or positive hepatitis C RNA test result at screening or within 3 months before the first dose of the study treatment unless the participant can meet the following criteria:

    * RNA test negative
    * Successful anti-viral treatment (usually 8 weeks duration) is required, followed by a negative hepatitis C virus RNA test after a washout period of at least 4 weeks.
16. Current corneal epithelial disease except for mild punctate keratopathy.

    * NOTE: Participants with mild punctate keratopathy are allowed. Mild (Grade 1) punctuate keratopathy is characterized by the appearance of only a few, if any, microcyst-like epithelial changes (MECs), as identified in the slit-lamp examination, with a low density (non-confluent), and predominantly (≥80%) located in the periphery of the cornea
17. Intolerance or contraindications to anti-viral prophylaxis.
18. Unable to tolerate antithrombotic prophylaxis.
19. AL amyloidosis (light chain amyloidosis), active POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal plasma proliferative disorder, skin changes) or active plasma cell leukemia at the time of screening.
20. Exhibiting clinical signs of or with known history of meningeal or central nervous system involvement by MM.
21. Known immediate or delayed hypersensitivity reaction or idiosyncratic reaction to drugs chemically related to belantamab mafodotin or any of the components of the study treatment.
22. Use of an investigational drug within 14 days or 5 half-lives (whichever is shorter) preceding the first dose of study drug.
23. Plasmapheresis within 7 days before the first dose of the study drug.
24. Participants with active small and/or large intestinal disease which is not adequately controlled with the appropriate treatment (e.g., uncontrolled diarrheal disease).
25. Participants with uncontrolled skin disease.
26. Participants with any condition causing hypophosphatemia, hypokalemia or hypomagnesemia which is refractory to electrolyte replacement.
27. Participants with previous administration of a gamma secretase inhibitor.
28. Participants with concomitant administration of a strong or moderate CYP3A4 inhibitor or inducer.
29. Any serious and/or unstable pre-existing medical, psychiatric disorder or other conditions (including lab abnormalities) that could interfere with participant's safety, obtaining informed consent or compliance to the study procedures.
30. Participant must not have received a live or live-attenuated vaccine within 30 days prior to first dose of belantamab mafodotin.
31. Participant should not use contact lenses while receiving belantamab mafodotin.
32. Because of the embryo-fetal risk of lenalidomide, all participants must adhere to the lenalidomide pregnancy prevention program applied in their region.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-07-14 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Part 1: Dose-Limiting Toxicity (DLT) | Up to 28 days
  The number (%) of participants with DLTs using the DLT evaluable population.
Part 1 and 2: Adverse Events (AEs) and Serious adverse events (SAEs) | Up to 4 years
  The number (%) of participants with AEs and SAEs using the DLT evaluable and Safety populations
Part 1 and 2: Ocular Toxicity | Up to 4 years
  The number (%) of participants with grade 2 or above KVA events
Part 2: Overall Response Rate (ORR) | Up to 4 years
  ORR as per International Myeloma Working Group (IMWG) by Investigator Assessment; defined as the percentage of participants with a confirmed Partial Response (PR), Very Good Partial Response (VGPR), Complete Response (CR) or stringent Complete Response sCR in the intent-to-treat (ITT) set.

SECONDARY OUTCOMES:
Part 1 and 2: Lenalidomide Relative Dose Intensity (RDI) | Up to 4 years
  The RDI is defined as the percentage of the total administered over the total planned lenalidomide dose.
Part 1 and 2: Nirogacestat Relative Dose Intensity (RDI) | Up to 4 years
  The RDI is defined as the percentage of the total administered over the total planned nirogacestat dose.
Part 1 and 2: Cumulative dose of bentalamab mafodotin | Up to 4 years
  Cumulative administered dose of belantamab mafodotin in combination with lenalidomide, dexamethasone and nirogacestat i.e., the total dose of belantamab mafodotin that was administered.
Part 1: Overall Response Rate (ORR) | Up to 4 years
  Overall Response Rate as per IMWG by Investigator Assessment
Part 1 and 2: Time To Response (TTR) | Up to 4 years
  TTR as per IMWG by Investigator Assessment (ITT population). TTR is defined as the time (in months) between the date of randomization and the first evidence of confirmed response (PR or better) for participants who achieve a response (i.e., confirmed PR or better).
Part 1 and 2: Duration of Response (DoR) | Up to 4 years
  DoR is defined as the time (months) from first evidence of confirmed PR or better until the earliest date of: documented disease progression (PD) per IMWG response criteria; or death due to PD among participants who achieved a response of PR or better. For alive and progression-free participants, data will be censored at the date of initiation of the subsequent line of treatment or at the last date of FU that the participant was known to be alive and progression-free.
Part 1 and 2: Complete Response Rate (CRR) | Up to 4 years
  CRR is defined as the percentage of participants with a confirmed CR or sCR. The denominator will be the total number of participants in each population and group respectively.
Part 1 and 2: Very Good Partial Response (VGPR) or better | Up to 4 years
  VGPR or better as per IMWG by Investigator Assessment (ITT population). VGPR or better rate is defined as the percentage of participants with a confirmed VGPR, CR or sCR. The denominator will be the total number of participants in each population and group respectively.
Part 1 and 2: Minimal Residual Disease (MRD) negative rate | Up to 4 years
  MRD negativity rate (ITT population); defined as the number (%) of participants who achieve MRD negativity (at or below the threshold of 10^-5), assessed via NGF. The denominator will be the total number of participants in each population and group respectively.
Part 1 and 2: Progression Free Survival (PFS) | Up to 4 years
  PFS as per IMWG by Investigator Assessment (ITT population, Safety population). PFS is defined as the time (in months) from randomization until the earliest date of documented PD per IMWG, or death due to any cause. For participants who neither progress nor die, the PFS will be censored at the date of their last adequate disease assessment. For participants who start a new anti-myeloma treatment, PFS will be censored at the date of the last adequate assessment before the start of the new treatment. For a randomized participant who does not have any post-baseline disease assessments and who has not died, PFS will be censored at the randomization date.
Part 1 and 2: Overall Survival (OS) | Up to 4 years
  OS is defined as the time from first dose/randomization until death due to any cause. If a participant is not known to have died, survival time will be censored at the date of last contact ("last known date alive").
Part 1 and 2: Abnormal ocular findings | Up to 4 years
  Number (%) of participants with abnormal ocular findings (on ophthalmic exam) (DLT evaluable population, Safety population).
Part 1 and 2:Pharmacokinetics (PK) Analysis | Up to 4 years
  Concentration-time data: linear and semi-logistic unique profiles of concentration-time and the mean and median profiles (as applicable) will be graphically represented for belantamab mafodotin. Belantamab mafodotin concentrations will be presented for each participant and summarized (as applicable) at each PK timepoint.
  Additionally, concentration-time and the mean and median profiles (as applicable) will be graphically represented for nirogacestat. Nirogacestat concentrations will be presented for each participant and summarized (as applicable) at each PK timepoint.
Part 1 and 2:Ocular symptoms and related impacts | Up to 4 years
  Number of participants with changes from baseline and proportion of participants with within-participant meaningful change in self reported ocular symptoms and related impacts as measured by the OSDI questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Evangelos Terpos, Prof, Principal Investigator — Department of Clinical Therapeutics, School of Medicine, National Kapodistrian University of Athens (NKUA)
Locations (2):
- Greece (2):
  - General Hospital of Athens "Alexandra", NKUA, Therapeutic Clinic, Athens
  - Anticancer Hospital of Thessaloniki "Theageneio", Thessaloniki

IPD SHARING:
Plan to Share IPD: No